CLINICAL TRIAL: NCT07184723
Title: Investigating Practice Patterns in Symptomatic Non-ruptured Abdominal Aortic Aneurysms (AAA) in Europe
Acronym: DETHINE
Status: Recruiting | Type: Observational
Sponsor: Wilhelminenspital Vienna (Other)
Responsible Party: Principal Investigator, Prim PD Dr Afshin Assadian, Head of Department, Wilhelminenspital Vienna
Other Study IDs: EK_24_063_VK
Record Dates: First submitted 2025-07-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-06

CONDITIONS: Symptomatic Non-ruptured Abdominal Aortic Aneurysms
Keywords: abdominal aortic aneurysm; symptomatic non-ruptured; vascular surgery; Europe
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Symptomatic non-ruptured abdominal aortic aneurysms (snrAAA) remain a clinical challenge due to limited evidence and heterogeneous definitions and management strategies. Unlike ruptured AAAs, snrAAA lack large-scale population-based studies, primarily due to inconsistent application of standardised medical classifications (e.g., ICD-10) and international variability in definitions, diagnostic approaches, and treatment protocols. Optimal diagnostic pathways, preoperative risk assessments, and treatment strategies remain poorly defined, with minimal guidance from existing guidelines.

This study aims to conduct a multinational cross-sectional online survey with optional retrospective validation to assess current opinions on an institutional scale regarding the definition and management of patients with snrAAA in Europe. All European vascular centres offering elective and emergency AAA repair are eligible to participate. Multiple survey entries from the same institution are not allowed. Centres are also invited to participate in a retrospective observational validation, reporting diagnostic and therapeutic details of their last five snrAAA cases.

ELIGIBILITY:
Inclusion Criteria:

- Last 5 patients (aged >18 years) treated at a participating centre for symptomatic non-ruptured AAA (or the last patients in the preceding 5 years if they have treated less than 5 patients in 5 years)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: European vascular centres offering elective and emergency AAA repair
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants that define non-ruptured symptomatic AAA on clinical symptoms alone assessed by the snrAAA Questionaire | From August 2024 to June 2026
  The objective of this study is to provide insights into current practice strategies in the definition, diagnosis, preoperative optimization, and surgical care of patients with non-ruptured symptomatic AAA in Europe.
  Primary outcome measures will be count and proportion.

SECONDARY OUTCOMES:
Number of participants where the stated practices align with actual treatment patterns assessed by the snrAAA Questionaire and electronic Case Report Form | From August 2024 to June 2026
  In order to validate the data collected on the institutional standard of care for symptomatic non-ruptured AAA cases, centres are kindly invited to participate in a retrospective observational analysis in which they are asked to report the diagnostic and therapeutic procedure of the last 5 patients treated at their institution for symptomatic non-ruptured AAA (or the last patients in the preceding 5 years if they have treated less than 5 patients in 5 years).
  Secondary outcome measures will be count and proportion.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Vascular and Endovascular Surgery, Clinic Ottakring, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided